CLINICAL TRIAL: NCT04729543
Title: Adoptive Therapy With TCR Gene-engineered T Cells to Treat Patients With MAGE-C2-positive Melanoma and Head and Neck Cancer
Brief Title: MAGE-C2 TCR T Cell Trial to Treat Melanoma and Head and Neck Cancer
Acronym: MC2TCR
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Ludwig Institute for Cancer Research (Other); Dutch Cancer Society (Other); Stichting Coolsingel Rotterdam grant (Unknown); Jan Ivo Stichting grant (Unknown)
Responsible Party: Principal Investigator, A.A.M. van der Veldt, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL69011.000.19
Record Dates: First submitted 2020-11-18; First posted 2021-01-28 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Melanoma; Melanoma, Uveal; Head and Neck Cancer
MeSH Terms: conditions — Melanoma; Uveal Melanoma; Head and Neck Neoplasms | interventions — Azacitidine; Valproic Acid; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adoptive therapy with autologous MC2 TCR T cells (Experimental): * Accelerated titration phase I design and a subsequent single arm phase II study
  * Prior to T cell transfer (day 0), patients will be treated with valproic acid (dose 50 mg/kg/d, 7d; days -9 to day -3) and 5' azacytidine (dose 75mg/m2/d, 7d; days -9 to day -3)
  * Phase I: patients will be treated with one single intravenous administration of MC2 TCR T cells at 5 different escalated doses of 5x10E7, 5x10E8, 5x10E9,1.0x10E10, and the total number of cultured TCR T cells (i.e., usually 1.0-5.0 x10E10 TCR T cells). MC2 TCR T cell infusions will be supported by low dose of IL-2 administrations (s.c. 5x10E5 IU/m2 2qd for 5 days)
  * T cells will be processed using IL-15 and IL-21 to generate young T cells
  Interventions: Biological: Adoptive therapy with autologous MC2 TCR T cells

INTERVENTIONS:
Biological: Adoptive therapy with autologous MC2 TCR T cells — Adoptive therapy with autologous MC2 TCR T cells combined with AZA/VP
  Other Names: 5' Azacytidine (AZA); Valproic acid (VP); Interleukin 2 (IL2)

SUMMARY:
Single-centre, first-in-man phase I/II trial to demonstrate safety and efficacy of MAGE-C2/HLA-A2 TCR T cells (MC2 TCR T cells) in advanced melanoma (MEL) and head-and-neck carcinoma (HNSCC).

DETAILED DESCRIPTION:
In this patient study, the investigators target the Cancer Germline Antigen (CGA) MAGE-C2 (MC2), and use T cells with a young phenotype. MC2 is highly expressed in melanoma (MEL) and head-and-neck squamous cell carcinoma (HNSSC), but not in healthy adult tissues. The investigators isolated MC2-specific TCRs from MEL patients who showed clinical responses following vaccination that were accompanied by significant frequencies of anti-MC2 CD8 T cells in blood and tumor without apparent side effects. Following extensive evaluation of in vitro anti-tumor and self-reactivities, the investigators have selected a TCR that recognizes the ALK epitope in the context of HLA-A2 for clinical development. Furthermore, preclinical studies showed that epigenetic pretreatment of tumor cells, but not normal cells, up-regulated MC2 gene expression and resulted in enhanced recognition of MC2 by the selected TCR. In parallel to the above studies, the investigators renewed their GMP protocol to process T cells, using stimulating antibodies and cytokines, to generate T cells with a young phenotype.

In the current phase I/II study, the investigators explore the safety and anti-tumor efficacy of T cells engineered with the selected TCR in patients with MC2-positive MEL and HNSSC. The study contains the following unique elements:

* CGA not targeted before by T cell therapy
* New T cell processing method to generate young T cells
* Pretreatment of patients with epigenetic drugs
* No chemotherapy prior to T cell infusion

Leads:

* Clinical PI: Astrid van der Veldt, MD, PhD
* Clinical logistics: Karlijn de Joode, MD
* T cell production: Monique de Beijer, PhD; and Cor Lamers, PhD
* Coordinator/Preclinical PI: prof. Reno Debets, PhD

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent;
2. Age ≥ 18 years;
3. One of the following three malignancies:

   * Previously treated for unresectable or metastatic cutaneous or mucosal melanoma for whom no standard treatment is available (anymore);
   * Metastatic uveal melanoma, progressing after standard of care therapy, if available;
   * R/M HSNCC for whom no standard treatment is available anymore;
4. Patients must be HLA-A2*0201 positive;
5. Primary tumor and/or metastasis (archival or fresh biopsy) is positive for MC2 (>5% of tumor cells) according to immunohistochemistry;
6. Measurable disease according to RECIST v1.1;
7. At least one lesion, suitable for sequential mandatory tumor biopsies;
8. ECOG performance status of 0 or 1. Life expectancy ≥ 12 weeks;
9. Patients with melanoma must have had objective evidence of disease progression while on or after standard systemic therapy. The last dose of prior therapy (e.g. anti- PD-1, chemotherapy) must have been received more than 4 weeks prior to the start of study treatment. For melanoma patients who are treated with BRAF- and MEK inhibitors, an interval of 2 weeks between discontinuation of BRAF- and MEK inhibition and start of study treatment is sufficient;
10. Patients with R/M HNSCC must have had objective evidence of disease progression and are ineligible for or unwilling to get platinum-based chemotherapy or for whom no standard treatment is available;
11. Patients of both genders must be willing to practice a highly effective method of birth control during treatment and for four months after receiving the preparative regimen;
12. Patients must meet the following laboratory values at the screening visit in the absence of growth factors and/or transfusion support:

Hematology:

* absolute neutrophil count greater than 1.5x10^9/L;
* platelet count greater than 75x10^9/L;
* hemoglobin greater than 5 mmol/L or 8.0 in g/dl;

Chemistry:

* serum ALAT/ASAT less than 3 times the upper limit of normal (ULN), unless patients have liver metastasis (<5 times ULN);
* serum creatinine < 1.5 ULN;
* total bilirubin ≤ 20 micromol/L, except in patients with Gilbert's Syndrome who must have a total bilirubin ≤ 50 micromol/L;

Serology:

* seronegative for HIV antibody;
* seronegative for hepatitis B antigen, and hepatitis C antibody;
* seronegative for lues.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from participation of this study:

1. presence of symptomatic brain metastasis. Note: subjects with symptomatic brain lesions who have been definitively treated with stereotactic radiation therapy, surgery, or gamma knife therapy are eligible;
2. Presence of active brain metastasis defined as new or progressive brain metastasis at the time of study entry. Note: subjects with treated or stable brain metastasis are eligible;
3. Presence of leptomeningeal metastasis;
4. Presence of malignant pleural effusion or ascites;
5. Systemic chronic steroid therapy (>10 mg/day prednisone or equivalent) or any other immunosuppressive therapy within 7 days prior to leukapheresis or 72 hours prior to infusion of the MC2 TCR T cells. Note: local steroids such as topical, inhaled, nasal and ophthalmic steroids are allowed;
6. Active, known or suspected autoimmune disease or a documented history of autoimmune disease. Note: subjects with vitiligo, controlled type 1 diabetes mellitus on stable insulin dose, residual autoimmune-related hypothyroidism only requiring hormone replacement or psoriasis not requiring systemic treatment are permitted;
7. Any active systemic infections, coagulation disorders or other active major medical illnesses, such as active autoimmune diseases requiring anti-TNF treatment;
8. History of myocardial infarction, cardial angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 6 months of enrollment;
9. AEs of previous treatment. Toxicities associated with prior systemic and non- systemic treatment must have recovered to a grade 1 or less. Patients may have undergone minor surgical procedures or palliative radiotherapy (for non-target lesions) within the past 4 weeks, as long as all toxicities have recovered to grade 1 or less;
10. Women who are pregnant or breastfeeding. A negative pregnancy test before inclusion in the trial is required for all women of child bearing age;
11. Use of any live vaccines against infectious diseases within the last 3 months;
12. Active infection requiring systemic antibiotic therapy at start of study treatment;
13. Prior allogenic bone marrow or solid organ transplant;
14. History of known hypersensitivity to any of the investigational drugs used in this study;
15. Malignant disease, other than being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to start of study treatment, completely resected basal cell and squamous cell skin cancers and any completely resected carcinoma in situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2027-10-20 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of MC2 TCR T cells | 1 year
  MTD is determined using an accelerated titration phase with T cell doses as described in treatment arm; AEs are recorded according to CTCAE 5.0
Objective anti-tumor responses of MC2 TCR T cells | 2 years
  Anti-tumor responses are recorded according to RECIST v1.1 using the MTD from outcome 1

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Result] Lamers CH, van Steenbergen-Langeveld S, van Brakel M, Groot-van Ruijven CM, van Elzakker PM, van Krimpen B, Sleijfer S, Debets R. T cell receptor-engineered T cells to treat solid tumors: T cell processing toward optimal T cell fitness. Hum Gene Ther Methods. 2014 Dec;25(6):345-57. doi: 10.1089/hgtb.2014.051. PMID 25423330
- [Result] Kunert A, van Brakel M, van Steenbergen-Langeveld S, da Silva M, Coulie PG, Lamers C, Sleijfer S, Debets R. MAGE-C2-Specific TCRs Combined with Epigenetic Drug-Enhanced Antigenicity Yield Robust and Tumor-Selective T Cell Responses. J Immunol. 2016 Sep 15;197(6):2541-52. doi: 10.4049/jimmunol.1502024. Epub 2016 Aug 3. PMID 27489285
- [Result] Kunert A, Obenaus M, Lamers CHJ, Blankenstein T, Debets R. T-cell Receptors for Clinical Therapy: In Vitro Assessment of Toxicity Risk. Clin Cancer Res. 2017 Oct 15;23(20):6012-6020. doi: 10.1158/1078-0432.CCR-17-1012. Epub 2017 Jun 23. PMID 28645940

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/43/NCT04729543/Prot_SAP_000.pdf